CLINICAL TRIAL: NCT06036381
Title: Spatial and Temporal Characterization of Gliomas Using Radiomic Analysis
Acronym: GLIO-RAD
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Collaborators: Indian Statistical Institute, Kolkata (Unknown)
Responsible Party: Principal Investigator, Dr Archya Dasgupta, Assistant Professor, Radiation Oncology, Tata Memorial Centre
Other Study IDs: 4146
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioma
Keywords: Glioma; Radiomics; Artificial Intelligence; Machine learning
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Radiomic analysis of imaging - MRI, PET, CT — Radiomic analysis of imaging will be undertaken as a standard of care to develop computational algorithms for patients treated in our institution.

SUMMARY:
Glioma are type of primary brain tumors arising within the substance of brain. Different type of gliomas are seen which are classified depending upon pathological examination and advanced molecular techniques, which help to determine the aggressiveness of the tumor and outcomes. Artificial intelligence uses advanced analytical process aided by computer which can be undertaken on the medical images. We plan to use artificial intelligence techniques to identify the abnormal areas within the brain representing tumor from the radiological images. Also, similar approach will be undertaken to classify gliomas with good or bad prognosis, to differentiate glioma from other type of brain tumors, and to detect response after treatment.

DETAILED DESCRIPTION:
In the proposed retrospective study, images (MRI, CT, or PET) undertaken as part of standard of care (pre-treatment, post-operative, response assessment, and surveillance) will be analyzed. The DMG database maintaining records of patients registered in TMC neuro-oncology DMG will be screened to identify the patients eligible for the study. With approximately 500-600 gliomas seen annually and approximately 80-100 patients/year having pre-treatment imaging, we expect a ceiling of 1000 patients during 2010-2022, which will be the maximum number of patients used for the analysis. All the images will be downloaded from the PACS applying anonymization filters, with clinical records extracted by review of electronic medical records and radiation plans. Imaging pre-processing will be done, which will include skull stripping and registration across different modalities (e.g., MRI and CT) or different sequences (e.g., T1C, T2W, ADC) will be done using rigid or deformable algorithms as suited best for the modality. Image segmentation to classify the region of interest will be done and verified individually by a neuro-radiologist or nuclear medicine physician as appropriate. The segmentations will be done to identify T1-contrast enhancing region (CE), non-enhancing regions (NE), and necrosis (NEC) guided by T1-C, T2W, and T2-FLAIR areas. The contours and the images will be resampled to a uniform resolution for different sequences or modalities (e.g., T2W/ ADC/ PET) to match either with the 3D sequence (e.g., FSPGR sequence) or available images with the least slice thickness. Subsequently, normalization techniques (e.g., histogram normalization/ Z-score normalization) will be undertaken within the individual images and across the entire dataset to account or image heterogeneity, including field strength for MRI and different image acquisition parameters. For auto segmentation, both supervised and unsupervised machine learning algorithms will be applied. For the supervised model, the entire database will be split into training and test cohorts for the model and application development, respectively. The effectiveness of the automated model will be tested using the dice similarity coefficient between manually segmentation regions and AI-based segments. For prognostication of gliomas, the next step will include feature extraction, which will consist of first-order (including shape, histogram), second-order or higher-order (e.g., different texture features like GLCM, GLDM, GLSZM, etc.), or deep learning techniques will be employed. Delta-radiomics will include temporal changes in the radiomic features from different time points for the same patient within the entire volume and individual regions. Subsequently, feature reduction and selection techniques like LASSO, recursive feature elimination will be used to shortlist the number of features depending on the sample size. The outputs will be decided based on the modeling defined for specific class problems (e.g., tumor vs. edema, recurrence vs. pseudo progression, outcomes, tumor region of interest vs. non-tumoral area) as obtained from the clinical information. Any class imbalance will be addressed using methods like random subset sampling or SMOTE analysis for data augmentation of the minority class. Machine learning algorithms like LDA, k-NN, SVM, random forest, AdaBoost, etc., will be applied singularly or in combination as an ensembled classifier to find the model with best performance. Deep learning classifiers will be used along with feature-based modeling and compared to test the classifier's applicability. Validation techniques like leave-one-out validation, k-fold validation, and split (into training and test cohort) will be used to assess the stability of the machine learning model. Radiomic analysis will be done by data scientist/ study investigators with expertise in data analytics. All segmentations will be done on open-source software like ITK snap (itksnap.org) or 3D Slicer (slicer.org). Feature extraction and modeling will be done using open-source software like Python (python.org). With continuous advancements in computational science, available newer analytical techniques and platforms will be applied as appropriate by collaborators from Indian Statistical Institute, Kolkata, Machine Intelligence Unit by sharing of the anonymized data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glioma or glioma-mimicking pathology with imaging available in TMC between January 2010 and December 2022.

Exclusion Criteria:

* Imaging done outside TMC.
* Motion artifacts or other artifacts causing image degradation.
* Size of tumor or region of interest < 1 cm in the largest dimension

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be according to the Inclusion and Exclusion Criteria . Study Includes vulnerable participants also. Minors (up to 18 years),Elderly
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Autosegmentation of tumor | 3 years
  The correlation of tumor region between manual segmentation and artificial intelligence-based autosegmentation model will be assessed using the Dice coefficient of similarity.
Prognostication of gliomas | 3 years
  Radiomic signature in prognostication of gliomas with estimation of progression-free survival and overall survival using Kaplan Meier plots and radiomics score-based nomograms.

SECONDARY OUTCOMES:
Response assessment in gliomas | 3 years
  Response assessment of gliomas using artificial intelligence model-based prediction and comparison with actual response (like radionecrosis, progression) using confusion matrices and estimation of parameters like sensitivity, specificity, accuracy, area under curve.
Differentiation of glioma from non-glioma histology | 3 years
  Use of radiomics model to differentiate gliomas from other brain tumors, with performance indices calculated using sensitivity, specificity, accuracy, area under curve.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. ARCHYA DASGUPTA, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No